CLINICAL TRIAL: NCT02184936
Title: Precise and Rapid Assessment of Collaterals Using Multi-phase CTA in the Triage of Patients With Acute Ischemic Stroke for IA Therapy
Brief Title: Measuring Collaterals With Multi-phase CT Angiography in Patients With Ischemic Stroke
Acronym: PRove-IT
Status: Completed | Type: Observational
Sponsor: Carol Kenney (Other)
Responsible Party: Sponsor-Investigator, Carol Kenney, Study co-ordinator, University of Calgary
Organization: University of Calgary (Other)
Other Study IDs: 24416
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Ischemic Stroke
Keywords: CT Angiography, CT Perfusion, Ischemic Stroke, Collaterals
MeSH Terms: conditions — Ischemic Stroke | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- acute ischemic stroke
  Interventions: Other: standard of care

INTERVENTIONS:
Other: standard of care

SUMMARY:
Treatment of acute ischemic stroke (AIS) is aimed at salvaging viable but ischemic brain by opening the occluded artery and restoring anterograde perfusion as quickly as possible. Time saved while making critical decisions correctly is vital in AIS management. Conventional angiography is invasive, resource intensive and not feasible as a fast diagnostic tool. Perfusion CT and MRI are both susceptible to patient motion, need trained personnel to process and take at least 10-30 min to acquire and interpret. The investigators have developed a new imaging tool, multi-phase CT Angiography (CTA), which generates multiple time resolved images of backfilling arteries beyond a blocked artery filled by collaterals.

Investigators seek to determine: i) if patients with AIS will have a differential clinical response to early recanalization based on collateral status assessed on multi-phase CTA, ii) if the extent to which collateral assessment on multi-phase CTA resembles perfusion CT in predicting which patients will have good clinical outcome with early recanalization, iii) Identify determinants of variability in native collateral status in patients with acute ischemic stroke.

Investigators hypothesize that patients with good and intermediate collaterals on multi-phase CTA achieve good clinical outcome with early recanalization (within 4 hours of baseline imaging); patients with poor collaterals do not do well even with early recanalization.

Prove-IT is a prospective multi-center hospital-based cohort study of 500 consecutive patients with acute ischemic stroke presenting within 12 hours of stroke symptom onset with evidence of intracranial occlusion on routine CTA over 3 years. Calgary and seven other comprehensive stroke centers will recruit patients into this study. Primary outcome is defined as a National Institute of Health Stroke Scale (NIHSS) score of 0 to 2 at 24 hours or an 8-point drop in NIHSS score from baseline to 24 hours. Secondary outcomes are a) 90-day modified Rankin Score (mRS) 0-2 or equal to the pre-stroke mRS; b) percent neurologic improvement comparing NIHSS at baseline to 24 hours; c) 90-day NIHSS score 0-2; d) infarct volume on 24 hour imaging and e) parenchymal intracerebral hemorrhage type 1 and 2 (ECASS II criteria) at 24 hrs.

Prove-IT looks to establish the ideal imaging selection tool for intra-arterial (IA) and thrombolysis decisions in the setting of AIS which is widely available, and can quickly and reliably detect salvageable brain.

ELIGIBILITY:
Inclusion Criteria:

1. Patient presenting to the emergency department with symptoms consistent with ischemic stroke.
2. Age > 18 yrs.
3. Baseline imaging including multi-phase CTA done within 12 hours of stroke symptom onset and initiated before recanalization therapy.
4. Evidence of a visible and symptomatic intracranial occlusion on baseline CT-angiography (intracranial ICA, M1 MCA segment +/- intracranial ICA, proximal M2 MCA).
5. Treatment with IV tPA and/or IA therapy.

Exclusion Criteria:

1. Intracranial hemorrhage (ICH) identified on baseline CT.
2. Previous moderate to large stroke in the ipsilesional hemisphere.
3. Modified Rankin Scale > 2 at baseline.
4. Unable to have CT-angio performed due to recent estimated creatinine clearance eCCr<60 ml/min, contrast allergy or other reasons.
5. Participation in another study that results in the patient receiving an investigational drug or therapy.
6. Any terminal illness (patient not expected to survive > 1 year).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke presenting within 12 hours of stroke symptom onset with evidence of intracranial occlusion on routine CTA.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2012-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Major neurological improvement at 24 hours | 24 hours post stroke onset
  defined as a NIHSS score of 0 to 2 at 24 hours or an 8-point drop in NIHSS score from baseline to 24 hours.

SECONDARY OUTCOMES:
90 day clinical outcome | 90 days
  1. 90-day modified Rankin Score (mRS) 0-2 or equal to the pre-stroke mRS
  2. Ordinal (shift) analysis across the mRS scale
percent neurologic improvement comparing NIHSS at baseline to 24 hours | 24 hours
90-day NIHSS score 0-2 | 90 days
Radiological outcome | 24 hours
  infarct volume on 24 hour imaging and parenchymal intracerebral hemorrhage type 1 and 2 (ECASS II criteria) at 24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Bijoy Menon, MD, Principal Investigator — University of Calgary, Calgary Stroke Program
Locations (2):
- Foothills Medical Centre, Calgary, Alberta, Canada
- Arcispedale Sant'Anna · Department of Neurology, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No
No individual participant date will be shared, overall data( anonymous) will be available and shared